CLINICAL TRIAL: NCT07227961
Title: Evaluating the Implementation, Utility, and Clinical Importance of the Patient-Reported Outcome Measure Information System (PROMIS) in Sarcoma Patients: A Multi-Centered Prospective Cohort Study
Brief Title: PROMIS and Mobility Evaluation in Sarcoma Patients
Status: Recruiting | Type: Observational
Sponsor: University of Calgary (Other)
Collaborators: University of Toronto (Other); Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: HREBA.CC-25-0017
Record Dates: First submitted 2025-11-04; First posted 2025-11-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: Sarcoma; Giant Cell Tumor of Bone
Keywords: Patient reported outcomes; PROMIS; TESS; Mobility; Recovery; Surgery; App; Digital health; Sarcoma
MeSH Terms: conditions — Sarcoma; Giant Cell Tumor of Bone; Alzheimer Disease | interventions — Surgical Procedures, Operative; Methods; Transurethral Resection of Bladder; Amputation, Surgical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sarcoma: Adult patients treated with surgery for bone and soft tissue sarcoma, and giant cell tumor of bone
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — Any type of surgery performed to remove the primary tumor including resection, amputation, and bone stabilization.
  Other Names: Operation; Procedure; Tumor resection; Amputation; Bone stabilization

SUMMARY:
The goal of this is to validate the Patient-Reported Outcomes Measurement Information System (PROMIS) in sarcoma patients undergoing surgery, and to evaluate a novel smartphone app for collecting mobility data. The goals of the study include to:

1. Validate PROMIS as a patient outcome measure in sarcoma
2. Assess the effectiveness of a novel app for administering questionnaires and collecting mobility metrics
3. Compare PROMIS scores and mobility metrics to better evaluate recovery trajectories after surgery

Participants will complete PROMIS questionnaires at regularly scheduled intervals using the smartphone app. Questionnaires will be completed pre-operatively and at 6 weeks, 12 weeks, 6 months, and 12 months post-operatively. Additionally, the app will passively track mobility metrics such as daily step count, stairs climbed, and gait parameters to compare with PROMIS scores.

DETAILED DESCRIPTION:
Background & Rationale:

Sarcoma is a rare form of bone and soft tissue cancer, making up about 1% of all adult cancers. Management typically involves radiation therapy, chemotherapy, and surgical resection, with or without limb reconstruction. The diagnosis, intensive treatment regimen, and surgery-induced deficits significantly impact patient quality of life and function.

Evaluating outcomes in sarcoma is challenging due to disease heterogeneity, complexity, and variation in surgical strategy. Patient-reported outcomes measures are crucial for evaluating treatment outcomes and facilitating patient-centered care. Traditional validated PROMs, like the Toronto Extremity Salvage Score (TESS), have significant ceiling effects. PROMIS assesses physical, mental, and social well-being using item response theory in a standardized manner for precise and sensitive measures. PROMIS was developed with oncology research considerations and has been validated in both orthopaedic and oncology populations. However, the significance of PROMIS in orthopaedic oncology is not well understood.

Assessing patient reported outcomes is limited by survey completion rates, particularly in the oncology patients who have multiple medical appointments and care teams. To address these challenges, our team has developed ACTIVATION (Activity Capture To Investigate Voluntary ActiviTy In Orthopaedic populatioNs), a smartphone application (app) tailored to musculoskeletal oncology. Unlike general fitness or commercial health applications, ACTIVATION passively captures mobility metrics and remotely administers PROMIS questionnaires. The continuous data collection aligns real-world mobility with clinical recovery timelines, offering a more precise view of patient outcomes.

The overall aim of this study is to validate PROMIS in sarcoma patients undergoing surgery, and to evaluate a novel smartphone app for questionnaire administration and collection of mobility data.

Hypothesis:

PROMIS and mobility metrics will provide a holistic and granular view of recovery trajectories, and the use of a novel smartphone application will improve patient engagement and data collection.

Aims:

1. Compare PROMIS to the current gold standard, the Toronto Extremity Salvage Score (TESS), in sarcoma
2. Determine the minimal clinically important difference (MCID) for PROMIS in sarcoma
3. Assess the feasibility and usability of an novel app for remote PROMIS and TESS administration, and mobility data collection
4. Correlate PROMIS and TESS scores with mobility metrics to define recovery trajectories
5. Identify demographic and socioeconomic factors that influence app engagement

Methods:

Recruitment and Sample Size: The investigator will recruit all eligible subjects identified by musculoskeletal oncology surgeons at the four study sites. The investigators anticipates enrolling approximately 800 sarcoma patients based on current surgical volumes and patient capture rates for collecting quality of life and functional data.

Data Collection:

Patients will be asked to download the ACTIVATION app on their smartphone and complete a demographic intake form. Clinical data will be obtained through the local electronic medical record. The TESS and PROMIS global health, self-efficacy, physical function, upper extremity function, and pain interference questionnaires will completed through the ACTIVATION app. Completion of these forms will be prompted via push notifications pre-operatively and at 6 weeks, 3 months, 6 months, and 12 months post-operative. Additionally, the app will passively collect mobility metrics from the smartphone operating system including step count, distance travelled, flights climbed, gait asymmetry, distinct activity periods (>10 minutes), and total time active. In patients who have a compatible smart watch, the investigators will also collect physiologic parameters including VO2 max, heart rate, and heart rate variability. At the end of study participation, two additional surveys will be administered. The survey will collect feedback about the overall efficacy of the app and assess participant phone carrying habits.

Statistical Analysis:

Longitudinal changes in PROMIS scores will be analyzed using linear mixed-effects models with time and patient-level covariates (e.g. age, sex, race, socioeconomic status) as fixed effects and patient as a random effect. Logistic regression will identify predictors of PROMIS completion. MCIDs for PROMIS domains will be calculated using an anchor-based method with the Global Rating of Change. The sensitivity of PROMIS will be compared to TESS using correlation coefficients, Bland-Altman plots, and linear regression models.

Mobility data will undergo principal component analysis to derive a composite index capturing the key features of interest. ROC curves will assess whether mobility changes predict meaningful changes in PROMIS scores. Additionally, subgroup analysis will be performed to determine if differences in recovery exist based on tumor location, type of surgery, and adjuvant cancer therapies. Missing data will be evaluated for randomness and addressed using multiple imputation or maximum likelihood estimation as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of bone sarcoma, soft tissue sarcoma, or giant cell tumor of bone
* Tumors located in the pelvis, lower extremities, or upper extremities
* Primary or recurrent disease
* Undergoing operative tumor resection, including limb salvage surgery and amputation
* Has an iPhone or Android phone
* Speaks English

Exclusion Criteria:

* Metastatic bone tumor
* Diagnosis of atypical lipomatous tumor or dermatofibrosarcoma protuberans
* Currently pregnant or planning pregnancy within 6 months
* Unwilling or unable to attend follow-up evaluations
* Cognitive or communication barriers that impede completion of questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will enrol patients under the care of a musculoskeletal oncology surgeon at Foothills Medical Centre (Calgary, AB, Canada), Mount Sinai Hospital (Toronto, ON, Canada), Mayo Clinic Arizona (Phoenix, AZ, United States), and Mayo Clinic Minnesota (Rochester, MN, United States).
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Step count | From enrolment to one year post-operative
  Number of steps
Distance travelled | From enrolment to 1 year post-operative
  Kilometers
Flights of stairs climbed | From enrolment to 1 year post-operative
  Number of flights climbed
Gait asymmetry | From enrolment to 1 year post-operative
  Percentage
Distinct activity periods | From enrolment to 1 year post-operative
  Number of distinct activity periods >10 minutes
Total time active | From enrolment to 1 year post-operative
  Minutes
PROMIS Global Health | From enrolment to 1 year post-operative
  Scored using standardized T-scores with a mean of 50 and a standard deviation of 10. Scores above 50 indicate more of the measured trait, while scores below 50 indicate less.
PROMIS Self Efficacy | From enrolment to 1 year post-operative
  Scored using standardized T-scores with a mean of 50 and a standard deviation of 10. Scores above 50 indicate more of the measured trait, while scores below 50 indicate less.
PROMIS Pain Interference | From enrolment to 1 year post-operative
  Scored using standardized T-scores with a mean of 50 and a standard deviation of 10. Scores above 50 indicate more of the measured trait, while scores below 50 indicate less.
PROMIS Physical Function | From enrolment to 1 year post-operative
  Scored using standardized T-scores with a mean of 50 and a standard deviation of 10. Scores above 50 indicate more of the measured trait, while scores below 50 indicate less.
PROMIS Upper Extremity Function | From enrolment to 1 year post-operative
  Scored using standardized T-scores with a mean of 50 and a standard deviation of 10. Scores above 50 indicate more of the measured trait, while scores below 50 indicate less.
Toronto Extremity Salvage Score Lower Extremity | From enrolment to 1 year post-operative
  Sum of patient responses for each question on a 5-point Likert scale, excluding "not applicable" items. The sum is then divided by the maximum possible score and multiplyed by 100 to yield a final score between 0 and 100. A score of 100 indicates no functional disability and 0 indicates the worst functional disability.
Toronto Extremity Salvage Score Upper Extremity | From enrolment to 1 year post-operative
  Sum of patient responses for each question on a 5-point Likert scale, excluding "not applicable" items. The sum is then divided by the maximum possible score and multiplyed by 100 to yield a final score between 0 and 100. A score of 100 indicates no functional disability and 0 indicates the worst functional disability.
Maximal oxygen consumption (VO2 max) | From enrolment to 1 year post-operative
  Litres per minute. A higher VO2 max indicates that the body is more efficient at using oxygen to produce energy in the muscles.
Heart rate | From enrolment to 1 year post-operative
  Beats per minute
Heart rate variability | From enrolment to 1 year post-operative
  Milliseconds. Measures the variation in time between each beat of your heart, with a higher score generally indicating better physical fitness.

SECONDARY OUTCOMES:
App Survey | Single collection time point at 1 year post-operative.
  Survey administered at the end of study participation to assess satisfaction and user-friendliness of the ACTIVATION app using Liekert scales. Survey also contains three short answer responses collecting feedback about the app and gathering data on technical difficulties. Last section of the survey contains questions about phone use habits using multiple choice questions..

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Rochester, Minnesota
- Canada (2):
  - Foothills Medical Centre, Arthur J Child Comprehensive Cancer Centre, University of Calgary, Calgary, Alberta
  - Mount Sinai Hospital, University of Toronto, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
To protect participant privacy and confidentiality, the investigators will not share IPD with other researchers. The study involves sensitive or identifiable health information and the consent obtained from participants does not include permission to share their individual-level data publicly or with third parties.

REFERENCES:
- [Background] Tyser AR, Beckmann J, Franklin JD, Cheng C, Hon SD, Wang A, Hung M. Evaluation of the PROMIS physical function computer adaptive test in the upper extremity. J Hand Surg Am. 2014 Oct;39(10):2047-2051.e4. doi: 10.1016/j.jhsa.2014.06.130. Epub 2014 Aug 16. PMID 25135249
- [Background] Hung M, Stuart AR, Higgins TF, Saltzman CL, Kubiak EN. Computerized Adaptive Testing Using the PROMIS Physical Function Item Bank Reduces Test Burden With Less Ceiling Effects Compared With the Short Musculoskeletal Function Assessment in Orthopaedic Trauma Patients. J Orthop Trauma. 2014 Aug;28(8):439-43. doi: 10.1097/BOT.0000000000000059. PMID 24378399
- [Background] Jensen RE, Potosky AL, Reeve BB, Hahn E, Cella D, Fries J, Smith AW, Keegan TH, Wu XC, Paddock L, Moinpour CM. Validation of the PROMIS physical function measures in a diverse US population-based cohort of cancer patients. Qual Life Res. 2015 Oct;24(10):2333-44. doi: 10.1007/s11136-015-0992-9. Epub 2015 May 3. PMID 25935353
- [Background] Blank AT, Lerman DM, Shaw S, Dadrass F, Zhang Y, Liu W, Hung M, Jones KB, Randall RL. PROMIS(R) scores in operative metastatic bone disease patients: A multicenter, prospective study. J Surg Oncol. 2018 Sep;118(3):532-535. doi: 10.1002/jso.25159. Epub 2018 Aug 16. PMID 30114336
- [Background] Garcia SF, Cella D, Clauser SB, Flynn KE, Lad T, Lai JS, Reeve BB, Smith AW, Stone AA, Weinfurt K. Standardizing patient-reported outcomes assessment in cancer clinical trials: a patient-reported outcomes measurement information system initiative. J Clin Oncol. 2007 Nov 10;25(32):5106-12. doi: 10.1200/JCO.2007.12.2341. PMID 17991929
- [Background] Ploetze KL, Dalton JF, Calfee RP, McDonald DJ, O'Keefe RJ, Cipriano CA. Patient-Reported Outcomes Measurement Information System physical function correlates with Toronto Extremity Salvage Score in an orthopaedic oncology population. J Orthop Translat. 2019 Mar 8;19:143-150. doi: 10.1016/j.jot.2019.02.004. eCollection 2019 Oct. PMID 31844622
- [Background] Ogura K, Uehara K, Akiyama T, Shinoda Y, Iwata S, Tsukushi S, Kobayashi E, Hirose T, Yonemoto T, Endo M, Tanzawa Y, Nakatani F, Kawano H, Tanaka S, Kawai A. Minimal clinically important differences in Toronto Extremity Salvage Score for patients with lower extremity sarcoma. J Orthop Sci. 2020 Mar;25(2):315-318. doi: 10.1016/j.jos.2019.03.022. Epub 2019 Apr 16. PMID 31000377
- [Background] Hassani M, Mate KKV, Turcotte R, Denis-Larocque G, Ghodsi E, Tsimicalis A, Goulding K. Uncovering the gaps: A systematic mixed studies review of quality of life measures in extremity soft tissue sarcoma. J Surg Oncol. 2023 Sep;128(3):430-437. doi: 10.1002/jso.27390. PMID 37537979
- [Background] Vijayakumar G, Blank AT. Patient-reported outcome tools in musculoskeletal oncology. J Surg Oncol. 2023 Sep;128(3):418-424. doi: 10.1002/jso.27386. PMID 37537983
- [Background] Goulding KA, Wilke BK, Kiernan HC, Houdek MT, Sherman CE. Skeletal Sarcomas: Diagnosis, Treatment, and Follow-up from the Orthopedic Oncologist Perspective. Radiol Clin North Am. 2022 Mar;60(2):193-203. doi: 10.1016/j.rcl.2021.11.001. PMID 35236588
- [Background] Gutowski CJ, Basu-Mallick A, Abraham JA. Management of Bone Sarcoma. Surg Clin North Am. 2016 Oct;96(5):1077-106. doi: 10.1016/j.suc.2016.06.002. PMID 27542644
- [Background] Walczak BE, Irwin RB. Sarcoma chemotherapy. J Am Acad Orthop Surg. 2013 Aug;21(8):480-91. doi: 10.5435/JAAOS-21-08-480. PMID 23908254
- [Background] Burningham Z, Hashibe M, Spector L, Schiffman JD. The epidemiology of sarcoma. Clin Sarcoma Res. 2012 Oct 4;2(1):14. doi: 10.1186/2045-3329-2-14. PMID 23036164

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-11-03): https://cdn.clinicaltrials.gov/large-docs/61/NCT07227961/Prot_SAP_000.pdf
  • Informed Consent Form (2025-11-03): https://cdn.clinicaltrials.gov/large-docs/61/NCT07227961/ICF_001.pdf